CLINICAL TRIAL: NCT05951634
Title: Clinical Investigation Plan (CIP) for: Safety and Performance Study for Arterial Large Hole Vascular Closure Device - ELITE Study
Brief Title: Safety and Performance Study for Arterial Large Hole Vascular Closure Device
Acronym: ELITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P935-00
Record Dates: First submitted 2023-06-29; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Large Hole Percutaneous Arterial Closure
Keywords: Arterial closure; Percutaneous arterial closure; Large hole arterial closure; Large bore arterial closure

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicentre, single-arm study to investigate the safety and efficacy of the PerQseal Elite.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Device Arm (PerQseal Elite) (Experimental): Large hole percutaneous arterial closure device - PerQseal Elite
  Interventions: Device: PerQseal ELITE

INTERVENTIONS:
Device: PerQseal ELITE — Percutaneous ELITE Arterial Closure Device
  The term PerQseal Elite used singularly refers to the closure system comprising the closure device and Introducer. These individually are referred to as: "PerQseal Elite VCD" or "PerQseal Elite closure device" and/or "PerQseal Elite Introducer".

SUMMARY:
To study will assess safety and performance of the PerQseal Elite Closure Device when used with the 18F PerQseal Elite Introducer to percutaneously close femoral artery punctures and to induce arterial haemostasis in patients undergoing endovascular procedures requiring an arteriotomy created by 14 to 22 F sheaths.

Note, for reference purposes, it is expected arteriotomies created with 14 to 22 F sheaths will create an arteriotomy in the range of 16 - 26 F (being the outer diameter of these sheaths).

DETAILED DESCRIPTION:
This study will be a prospective, multi-centred, non-randomized study to investigate the safety and performance of the PerQseal Elite. The study shall not be blinded prior to, during or post the procedure. All patients undergoing an endovascular procedure requiring an arteriotomy created by 14 to 22 F sheaths, via the common femoral artery will be screened against the inclusion/exclusion criteria.

All subjects shall have a pre-discharge, 30-Days ± 7-Days and 180-Days ± 30-Days follow-up assessment. All safety data from the study will be assessed by the Data Safety Monitoring Committee on a continuous basis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years.
2. Clinically indicated for a percutaneous arterial interventional catheter-based procedure, e.g., transcatheter aortic valve replacement/implantation (TAVR/TAVI) or endovascular abdominal aortic aneurysm repair (EVAR), or thoracic endovascular aortic aneurysm repair (TEVAR), or use of a circulatory assist device or extracorporeal oxygenation using a common femoral arteriotomy created by a 14 to 22F sheath (arteriotomy up to 26F).
3. Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
4. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.

Exclusion Criteria:

Baseline Exclusion Criteria:

1. Evidence of current systemic bacterial or cutaneous infection, including groin infection,
2. Known bleeding diathesis, definite or potential coagulopathy, platelet count < 100,000/µl or subjects on long term anticoagulants with an INR > 2 within 12 hours prior to index procedure,
3. Significant anaemia (example: haemoglobin < 9 g/dL or haematocrit < 27%), within 24 hours prior to index procedure,
4. Known type II heparin-induced thrombocytopenia,
5. Documented left ventricular ejection fraction < 20%,
6. Ipsilateral or contralateral lower extremity amputation,
7. Previous groin surgery within the region of the ipsilateral access,
8. Claudication (Rutherford category 3 or greater), documented untreated iliac or common femoral artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of target leg,
9. Known existing nerve damage in the target leg,
10. Renal insufficiency (Glomerular Filtration Rate ≤ 30 ml/min or baseline serum creatinine > 2.5 mg/dl) or on renal replacement therapy,
11. Known allergy to any of the materials used in the PerQseal Elite device (refer to Investigator's Brochure),
12. Subject is unsuitable for surgical repair of the target leg access site,
13. Subject has undergone a percutaneous procedure greater than 8F sheath in the target leg, within the 90-days prior to index procedure,
14. Subject has undergone a percutaneous procedure of 8F sheath or less using an absorbable intravascular closure device for haemostasis, in the target leg, within the 90-days prior to index procedure,
15. Subject has undergone a percutaneous procedure of 8F sheath or less using a suture mediated closure device or manual/mechanical pressure for haemostasis in the target leg, within the 30-days prior to index procedure,
16. Evidence of marked tortuosity of the femoral or external iliac arteries in the target leg, based on pre-primary procedure CT angiography,
17. Evidence of arterial diameter stenosis > 20% within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
18. Evidence of anterior wall calcification of the target common femoral artery (other than small, diffuse deposits which in the opinion of the investigator will not impede the vascular closure procedure) within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
19. Target femoral artery diameter is less than 7 mm, based on pre-primary procedure CT angiography,
20. Further planned endovascular/catheter-based procedure in the target leg in the 30-days following the index procedure,
21. Subject is enrolled in another investigational medical device or drug study,
22. Subject has been previously enrolled in this clinical study,
23. Current COVID-19 infection (with or without symptoms), recent positive test for COVID-19 within two weeks, or recent exposure to a person with COVID-19 infection within two weeks.

    Procedural Exclusion Criteria:* If any Procedural Exclusion Criteria listed below are met, then closure with PerQseal Elite device is not permitted,
24. Initial common femoral arterial access achieved with manual palpation or blind arterial stick access, without use of an image guided approach (ultrasound or angiography),
25. Difficult dilation during initial target femoral artery access (e.g., that damages or kinks dilators) while step-dilating up to the large-bore device,
26. During arterial puncture, the target femoral artery suspected to have experienced a posterior arterial wall needle puncture or underwent > one needle puncture during the primary procedure, with a needle larger than a micropuncture needle (> 21 gauge or > 0.819 mm diameter). (Note: not an exclusion if micropuncture technique under ultrasound guidance used for femoral artery access [Ref. 19, 20]),
27. Subject has a tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than 8 cm,
28. Significant blood loss requiring transfusion of blood products during primary procedure or within 30-days prior to index procedure,
29. Activated clotting time (ACT) > 300 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 300 seconds for more than 24 hours after index procedure,
30. Target puncture site is in a vascular graft,
31. Target arteriotomy greater than 26F,
32. Target arteriotomy in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 15 mm proximal of the bifurcation of the superficial femoral/ profunda femoris artery, (apex of bifurcation overlying the femoral head),
33. Target arteriotomy located at the level or above the inferior epigastric artery and/or beneath or above the inguinal ligament based on bony/arterial landmarks (above femoral head on A-P projection),
34. Subjects with an acute haematoma > 4 cm diameter, arteriovenous fistula, pseudoaneurysm or intraluminal thrombosis at the target access site identified intra-procedurally,
35. Evidence of bleeding around the primary procedure sheath (VARC type 1/BARC type 2 or higher),
36. Intra-procedural angiographic evidence of arterial laceration, dissection or stenosis within the femoral artery that would preclude use of the PerQseal Elite device,
37. Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) at the time of planned vascular closure,
38. Systolic blood pressure < 90 mmHg at the time of planned vascular closure. *May not be known until after the patient has given informed consent and the procedure has started. In this event, the PerQseal Elite should not be used and the patient should be considered excluded from the study and intention to treat analysis.

Note: The use of a secondary closure device in the same leg is prohibited during this study. A note to this effect should be entered into the patient's medical records.

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Major access site complications | through 30 Days
  Rate of major access site complications attributable to the PerQseal Elite device
Primary Effectiveness Endpoint - Time to Haemostasis | 20 Minutes
  Time to Haemostasis (TTH) defined as elapsed time in minutes from PerQseal Elite (Introducer-sheath and Delivery-device) removal to first observed cessation of common femoral artery (CFA) bleeding, excluding cutaneous or subcutaneous oozing, and in the absence of a developing haematoma.

SECONDARY OUTCOMES:
Secondary Safety Endpoint - Incidence of Minor Access Site Complications | Through 30 Days
  The Incidence of minor access site complications attributable to the PerQseal Elite device
Secondary Effectiveness Endpoint - PerQseal Elite Technical Success Rate | 10 Minutes
  Defined as the number of PerQseal Elite devices that are deployed and achieve haemostasis (i.e., cessation of arterial bleeding excluding cutaneous or subcutaneous oozing) without need for more than 10 minutes of firm, adjunctive manual compression or alternative treatment (other than adjunctive endovascular ballooning) at target access site, divided by the total number of PerQseal Elite devices where deployment was attempted, within the mITT population
Secondary Effectiveness Endpoint - PerQseal Elite Treatment Success Rate | through 30 days
  Defined as the number of subjects who meet PerQseal Elite Technical Success without experiencing a device related Major Access Site Complication (based on CEC adjudication) through 30-days, divided by the total number of subjects where PerQseal Elite device deployment was attempted, within the mITT population.
Secondary Effectiveness Endpoint - Time to Device Deployment | 20 Minutes
  Defined as the time from insertion of the PerQseal Elite delivery device into the PerQseal Elite Introducer sheath to complete removal of the PerQseal Elite (delivery device and introducer-sheath) from the subject following PerQseal Elite deployment.
Secondary Effectiveness Endpoint - Time to Ambulation | through 24 hours
  Defined as the elapsed time from PerQseal Elite removal from the subject post deployment until the subject can walk 20 feet/6 meters without arterial re-bleeding at the target access site. This endpoint will be evaluated only for subjects who are ambulatory (e.g., not confined to wheelchair or bed) at the time of enrolment.
Secondary Effectiveness Endpoint - Total Closure Time | 40 Minutes
  Total Closure Time is defined as: Time to Haemostasis (TTH) plus Time to Device Deployment (TTDD).

IPD SHARING:
Plan to Share IPD: No